CLINICAL TRIAL: NCT04820504
Title: Augmented Infant Resuscitator (AIR): Transitioning a Novel Behavior Change Innovation to Drive Newborn Ventilation Skills Enhancement
Brief Title: Augmented Infant Resuscitator to Enhance Newborn Ventilation
Acronym: AIR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Kristian R. Olson, M.D., Associate Professor, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2013P002204
Record Dates: First submitted 2021-02-17; First posted 2021-03-29 (Actual); Last update posted 2021-03-29 (Actual); Status verified 2021-03

CONDITIONS: Asphyxia Neonatorum; Birth Asphyxia; Perinatal Asphyxia
MeSH Terms: conditions — Asphyxia Neonatorum

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Blinded to visual feedback from AIR device (Placebo Comparator): Providers did not receive AIR device feedback during newborn mannequin ventilation
  Interventions: Device: AIR device without feedback
- Not blinded to visual feedback from AIR device (Experimental): Providers did receive AIR device feedback during newborn mannequin ventilation
  Interventions: Device: Augmented Infant Resuscitator (AIR)

INTERVENTIONS:
Device: Augmented Infant Resuscitator (AIR) — Device provides visual feedback related to air leak, obstruction, hyperventilation, hypoventilation, and harsh breaths
  Other Names: AIR device with feedback
  Arms: Not blinded to visual feedback from AIR device
Device: AIR device without feedback — Device provides no visual feedback to clinician but records data on ventilation effectiveness
  Arms: Blinded to visual feedback from AIR device

SUMMARY:
Augmented Infant Resuscitator (AIR) is an inexpensive add-on, compatible with nearly every existing bag-valve mask and many types of ventilation equipment. AIR monitors ventilation quality and provides real-time objective feedback and actionable cues to clinicians to both shorten training times and improve resuscitation quality, adoption, retention, and confidence.

DETAILED DESCRIPTION:
Longitudinal, randomized control trial that examined the effectiveness of AIR among 270 participants, with 1,080 recorded ventilation scenarios, and across 20 sites in Uganda and the U.S. Birth attendants - including a mix of midwives, nurses, respiratory therapists, pediatricians, and neonatologists - with recent HBB and/or NRP training were recruited to participate in this randomized control trial. Participants ventilated training mannequins for a fixed duration of time. Participants were randomized to receive visual feedback from AIR (intervention) or have the AIR feedback covered (control). They were then requested to administer effective ventilation and verbally assess the mannequin condition. All mannequins appeared to be identical, but each session's mannequin was randomly selected with an upper airway that was normal, partially leaking, or partially obstructed.

ELIGIBILITY:
Inclusion Criteria:

* Midwives, nurses, respiratory therapists, pediatricians, and neonatologists working as birth attendants in select hospitals in Uganda and the U.S. who are either previous trained in Helping Babies Breathe (HBB) and/or have a current Newborn Resuscitation Program (NRP) certification.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2016-11-01 (Actual); Study Completion 2016-11-01 (Actual)

PRIMARY OUTCOMES:
Effective bag-mask ventilation | 2 minutes
  Duration of effective bag-mask ventilation by clinician during a 2-minute trial. [This will be a cumulative duration of the two minutes. This is measured internally from the AIR device. "Effective ventilation" is defined as having all three of the following conditions simultaneously: (1) Correct rate (30-60 breaths per minute); (2) Absence of significant leak (compliance >4.0mL/cm H2O); and (3) Absence of a significant airway blockage (defined as compliance <0.10 mL/cm H2O or resistance >90 cmH2O/L/s). These measurements are determined by sensors in the AIR device for both arms of the study. Their accuracy for manikin use was determined to be 100% in the following trial: Bennett el al. Anesth Analgesia. 2018 Mar;126(3):947-955. doi: 10.1213/ANE.0000000000002432.]
Time to effective bag-mask ventilation | 2 minutes
  How long it takes for clinician to achieve effective ventilation during 2-minute trial. [This is time from when the mask first touches the face of the manikin until all three icons are green. This is measured by a Research Assistant using a stop-watch. Again, "Effective ventilation" is defined as having all three of the following conditions simultaneously and is indicated to the RA by all three icons on the AIR device turning green: (1) Correct rate (30-60 breaths per minute); (2) Absence of significant leak (compliance >4.0mL/cm H2O); and (3) Absence of a significant airway blockage (defined as compliance <0.10 mL/cm H2O or resistance >90 cmH2O/L/s). These measurements are determined by sensors in the AIR device for both arms of the study. Their accuracy for manikin use was determined to be 100% in the following trial: Bennett et al. Anesth Analgesia 2018 Mar;126(3):947-955. doi: 10.1213/ANE.0000000000002432.]
Clinician's correct assessment of mannequin airway issues | 2 minutes
  Ability of clinician to correctly assess three different manikin airway issues: normal, air leak, or obstruction. [Manikin "conditions" are blinded to the participants and were either normal (as supplied by the manufacturer, had a "leak" insert (introduced compliance >4mL/cm H2O), or had an "obstruction" insert (introduced a reduction in compliance <0.10mL/cm H2O and resistance >90 cm H2O/L/s. As per the parameters in the following paper: Bennett et al. Anesth Analgesia. 2018 Mar;126(3):947-955. doi: 10.1213/ANE.0000000000002432.]

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bennett DJ, Itagaki T, Chenelle CT, Bittner EA, Kacmarek RM. Evaluation of the Augmented Infant Resuscitator: A Monitoring Device for Neonatal Bag-Valve-Mask Resuscitation. Anesth Analg. 2018 Mar;126(3):947-955. doi: 10.1213/ANE.0000000000002432. PMID 28863023
- [Derived] Data S, Nelson BD, Cedrone K, Mwebesa W, Engol S, Nsiimenta N, Olson KR. Real-Time Digital Feedback Device and Simulated Newborn Ventilation Quality. Pediatrics. 2023 Nov 1;152(5):e2022060599. doi: 10.1542/peds.2022-060599. PMID 37873596